CLINICAL TRIAL: NCT06475651
Title: Characterization and Contribution of Genome-wide DNA Methylation (DNA Methylation Episignatures) in Rare Diseases With Prenatal Onset
Acronym: FOETEPISIGN
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231311
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Rare Fetal Genetic Diseases; Congenital Malformation
Keywords: Congenital malformation; DNA methylation abnormalities; Episignature; CHD7 gene; KMT2D gene; HYLS1 gene; TCTN3 gene; FLVCR2 gene; CHARGE syndrome; KABUKI syndrome
MeSH Terms: conditions — Congenital Abnormalities; CHARGE Syndrome; Hydrolethalus Syndrome 1; Kabuki syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — All the biological tissues required to carry out this pilot study (lung, blood, amniotic fluid and extracted DNA) come from a biological collection already constituted and declared as part of the diagnosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Workpackage 1, group 1: Patients (children) with CHARGE syndrome
  Interventions: Genetic: Methylation analysis
- Workpackage 1, group 2: Healthy negative controls (children) matched for age and sex
  Interventions: Genetic: Methylation analysis
- Workpackage 1, group 3: Fetuses with CHARGE syndrome
  Interventions: Genetic: Methylation analysis
- Workpackage 1, group 4: Fetuses with no genetic pathology
  Interventions: Genetic: Methylation analysis
- Workpackage 2, group 5: Patients (children) with KABUKI syndrome
  Interventions: Genetic: Methylation analysis
- Workpackage 2, group 6: Fetuses with KABUKI syndrome
  Interventions: Genetic: Methylation analysis
- Workpackage 3, group 7: Fetuses with hydrolethalus syndrome
  Interventions: Genetic: Methylation analysis
- Workpackage 3, group 8: Fetuses with Meckel/OFD IV syndrome
  Interventions: Genetic: Methylation analysis
- Workpackage 3, group 9: Fetuses with Fowler syndrome
  Interventions: Genetic: Methylation analysis

INTERVENTIONS:
Genetic: Methylation analysis — Genomic DNA will be treated with bisulfite. 500 ng of processed DNA is then hybrized on an EPICv2 array Infinium methylation (Illumina, San Diego, CA, USA). This microarray enables the analysis of approximately 865 000 methylation sites at promoters, enhancers, CpG islands, intergenic and intragenic regions. It is the most widely used chip in the literature, including almost all of the EPIGENETIC SIGNATURES reported in human pathology.

SUMMARY:
It is necessary to define reference DNA Methylation Episignatures from fetal DNA. The hypotheses are:

* It is possible to define reference DNA Methylation Episignatures from fetal DNA extracted from amniotic fluid or frozen tissues collected during the postmortem examination
* Fetal DNA Methylation Episignatures may be different to postanal DNA Methylation Episignatures defined on DNA extracted from blood

DETAILED DESCRIPTION:
Congenital anomalies (CA) complicate 3 to 5% of pregnancies and may be associated with genetic disorders. Diagnosis of genetic diseases is a major medical challenge, especially during pregnancy.

Over the past two decades, next-generation sequencing (NGS) has revolutionized our ability to identify the genetic condition associated with CA. During pregnancy, prenatal exome sequencing identified an additional diagnosis in around 30% of fetuses with CA when standard chromosomal investigations (karyotype and chromosomal microarray analysis, CMA) fail to provide a diagnosis.

Despite these major advances, around 40% of rare diseases remain unsolved, including 10-15% of patients harboring variants of uncertain significance (VUS).

After birth, additional functional analyses ("multi-OMICS"), including genome-wide DNA methylation studies, may be offered to reclassify VUS.

DNA methylation anomalies play an important role in pathologies (developmental disorders and oncology).

DNA methylation Episignatures, defined as the cumulative DNA methylation patterns occurring at multiple CpG dinucleotides across the genome, have been recognized to be intricately associated with many human traits, including age, sex, and disease status. Recently, DNA Methylation Episignatures have been identified in the blood of children or adults for several well-characterized genetic diseases. However, these postnatal DNA Methylation Episignatures cannot be used during pregnancy, because DNA methylation changes from one tissue to another and during time, especially during fetal developpement. In addition, the tissues available during pregnancy are different from those analyzed postnatally (blood).

ELIGIBILITY:
Inclusion Criteria:

* Patient Inclusion Criteria:

  * Fetuses with a postmortem examination as part of the etiological diagnosis of developmental abnormality within the Genomic Medicine of Rare Diseases department of the Necker Children's Hospital, and whose DNA extracted from lung and amniotic fluid is available
  * OR a child cared for in the Genomic Medicine for Rare Diseases department of the Necker Children's Hospital, and whose DNA extracted from whole blood is available
  * with pathogenic or probably pathogenic variation in a gene following CHD7, KMT2D, HYLS1, TCTN3 or FLVCR2
  * whose parents have consented to molecular genetic testing as part of diagnosis and research
* Negative Controls :

  * Fetuses with a postmortem examination as part of the etiological diagnosis of developmental abnormality within the Genomic Medicine of Rare Diseases department of the Necker Children's Hospital, and whose DNA extracted from lung and amniotic fluid are available
  * OR a child cared for in the Genomic Medicine for Rare Diseases department of the Necker Children's Hospital, and whose DNA extracted from whole blood is available
  * does not have pathogenic or probably pathogenic variation in a gene following CHD7, KMT2D, HYLS1, TCTN3 or FLVCR2
  * whose parents have consented to molecular genetic testing as part of diagnosis and research
* For everyone:

  • For living participants: Non-objection by holders of parental authority to the reuse of clinical data and biological samples collected and stored in the context of care (consent of care).

  • For deceased participants:
* Consent of the holders of parental authority to the use of the samples kept for research purposes, signed as part of the treatment
* No mention of opposition to the reuse of clinical data from the treatment in the patient's medical record

Exclusion Criteria:

* Refusal of postmortem examination in case of fetal loss
* Parents' refusal of molecular investigations

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population is derived from the Department of Genomic Medicine for Rare Diseases and the Multidisciplinary Center for Prenatal Diagnosis of the Necker-Enfants malades Hospital - APHP - GHU Paris Cité.
  The parents signed a consent to the storage and use of biological samples, stating that these samples taken as part of the treatment could be reused for medical research.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Epigenetic signature associated with pathogenic variations in the CHD7 gene (CHARGE Syndrome) | 12 months
  Evidence of epigenetic signature from fetal tissue DNA in fetuses with pathogenic or probably pathogenic variation
Epigenetic signature associated with pathogenic variations in the KMT2D gene (KABUKI syndrome) | 12 months
  Evidence of epigenetic signature from fetal tissue DNA in fetuses with pathogenic or probably pathogenic variation

SECONDARY OUTCOMES:
Differential methylation between fetal and postnatal epigenetic signature | 12 months
  Evidence of differential methylation between fetal an postnatal epigenetic signature
Differential methylation between tissue and amniotic fluid epigenetic signatures | 12 months
  Evidence of differential methylation between tissue and amniotic fluid epigenetic signatures
Statistical prediction parameter for each epigenetic signature | 12 months
  Measurement of the statistical prediction parameter for each epigenetic signature
Identification of a new epigenetic signature in foetal pathologies | 12 months
  Identification of news epigenetic signatures of exclusively pathologies associated with the HYLS1, TCTN3 and FLVCR2 genes

CONTACTS AND LOCATIONS:
Overall Officials: Manon TESSIER, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Department of Genomic Medicine for Rare Diseases and the Multidisciplinary Center for Prenatal Diagnosis of the Necker-Enfants malades Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Butcher DT, Cytrynbaum C, Turinsky AL, Siu MT, Inbar-Feigenberg M, Mendoza-Londono R, Chitayat D, Walker S, Machado J, Caluseriu O, Dupuis L, Grafodatskaya D, Reardon W, Gilbert-Dussardier B, Verloes A, Bilan F, Milunsky JM, Basran R, Papsin B, Stockley TL, Scherer SW, Choufani S, Brudno M, Weksberg R. CHARGE and Kabuki Syndromes: Gene-Specific DNA Methylation Signatures Identify Epigenetic Mechanisms Linking These Clinically Overlapping Conditions. Am J Hum Genet. 2017 May 4;100(5):773-788. doi: 10.1016/j.ajhg.2017.04.004. PMID 28475860
- [Background] Aref-Eshghi E, Kerkhof J, Pedro VP; Groupe DI France; Barat-Houari M, Ruiz-Pallares N, Andrau JC, Lacombe D, Van-Gils J, Fergelot P, Dubourg C, Cormier-Daire V, Rondeau S, Lecoquierre F, Saugier-Veber P, Nicolas G, Lesca G, Chatron N, Sanlaville D, Vitobello A, Faivre L, Thauvin-Robinet C, Laumonnier F, Raynaud M, Alders M, Mannens M, Henneman P, Hennekam RC, Velasco G, Francastel C, Ulveling D, Ciolfi A, Pizzi S, Tartaglia M, Heide S, Heron D, Mignot C, Keren B, Whalen S, Afenjar A, Bienvenu T, Campeau PM, Rousseau J, Levy MA, Brick L, Kozenko M, Balci TB, Siu VM, Stuart A, Kadour M, Masters J, Takano K, Kleefstra T, de Leeuw N, Field M, Shaw M, Gecz J, Ainsworth PJ, Lin H, Rodenhiser DI, Friez MJ, Tedder M, Lee JA, DuPont BR, Stevenson RE, Skinner SA, Schwartz CE, Genevieve D, Sadikovic B. Evaluation of DNA Methylation Episignatures for Diagnosis and Phenotype Correlations in 42 Mendelian Neurodevelopmental Disorders. Am J Hum Genet. 2020 Mar 5;106(3):356-370. doi: 10.1016/j.ajhg.2020.01.019. Epub 2020 Feb 27. PMID 32109418